CLINICAL TRIAL: NCT01738815
Title: Impact of Valproate on Angiogenesis and Histone Deacetylation in Bladder Cancer
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: State University of New York - Upstate Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 256549
Record Dates: First submitted 2012-11-28; First posted 2012-11-30 (Estimated); Last update posted 2021-10-22 (Actual); Status verified 2021-10

CONDITIONS: Hematuria; Bladder Cancer
Keywords: bladder cancer; hematuria; sodium valproate; valproic acid
MeSH Terms: conditions — Hematuria; Urinary Bladder Neoplasms | interventions — Valproic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- valproic acid (Experimental): Patients will be administered valproic acid (Depakote ER) for up to 30 days prior to tumor resection
  Interventions: Drug: Valproic Acid

INTERVENTIONS:
Drug: Valproic Acid — 500 mg orally, once daily for up to 30 days
  Other Names: Depakote ER

SUMMARY:
The goal of this study is to test whether the drug valproic acid can cause changes in bladder tumors that might inhibit their growth.

DETAILED DESCRIPTION:
Bladder cancer is the fourth most common cancer in the United States with over 60,000 new cases each year. It can usually be treated initially by insertion of an endoscope into the bladder and surgically removing the tumor, a procedure known as cystoscopy and trans-urethral resection of bladder tumor (TURBT). For most patients this procedure will successfully remove all of the detectable tumor. Unfortunately over 40% of all patients will develop a cancer recurrence in less than two years and all patients remain at increased risk of recurrence for the remainder of their lives. This risk requires life long monitoring and this is best accomplished with regular cystoscopic examinations. The goal of this study is to test whether the drug valproic acid can cause changes in bladder tumors that might inhibit their growth. Patients with suspected bladder cancer will be invited to participate in the study, if a tumor is observed during cystoscopy it will be sampled for research purposes and then according to standards of care, the patient scheduled for TURBT under general anesthesia. In the interval between discovery of a bladder tumor and resection, usually two to four weeks, the patient will be given valproic acid to take orally. In addition, tumors from patients with known or suspected bladder cancer referred for TURBT or cystectomy will be sampled. The tumor pieces obtained before and after taking valproic acid and from the referral patients not treated with valproic acid will be analyzed to see if the drug has changed what genes are active. We have found that valproic acid causes bladder cancer cells to make more of the protein, thrombospondin-1. This protein inhibits the growth of new blood vessels and so increased thrombospondin-1 in bladder tumors should inhibit their growth by decreasing the blood supply. Valproic acid may change thrombospondin-1 levels through inhibition of histone deacetylases. We will also assay HDAC activity in the tumor specimens. If valproic acid alters thrombospondin-1 levels and HDAC activity in bladder cancer patients further study to see if it can reduce growth will be justified. Valproic acid is a drug approved for the treatment of seizure disorders that is generally well tolerated with few side effects. It may prove useful in reducing bladder cancer recurrence and progression.

ELIGIBILITY:
Inclusion Criteria:

1. Patient over the age of 21
2. Bladder tumor suspected or confirmed
3. ECOG status 0 to 2
4. Premedication Lab values:

Absolute Neutrophil Count >750 cells/m3 AST/ALT less than 1.5xN Amylase less than 1.5xN Platelet Count > 125,000 PT/PTT > 1.3xN Hemoglobin > 8gm/dL Creatinine less than 1.5xN

Exclusion Criteria:

1. Allergy to valproic acid
2. Concurrent chemotherapy
3. Pre-menopausal women
4. Active systemic infection (HepatitisB,C)
5. Coagulation disorders
6. Concurrent medication: Tolbutamide, Warfarin, Zidovudine, Benzodiazepine, Clonazepam, Diazepam, Any anti-convulsant therapy
7. Seizure disorder
8. Dementia
9. History of Pancreatitis
10. HIV diagnosis/treatment
11. Liver disease/dysfunction

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2011-12 (Actual); Primary Completion 2013-05 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Thrombospondin-1 gene expression | 1 day
  Expression of thrombospondin-1 will be assayed using quantitative real-time PCR and western blotting. Comparisons will be intra-patient for paired specimens acquired prior to and after treatment and inter-patient for treated and un-treated patients.

SECONDARY OUTCOMES:
Angiogenesis, proliferation, and histone deacetylase activity markers | 1 day
  Histone deacetylase activity, angiogenesis, and proliferation markers will be assayed using qPCR and western blotting of tumor biopsy specimens. Comparisons will be intra-patient for paired specimens acquired prior to and after treatment and inter-patient for treated and un-treated patients.

CONTACTS AND LOCATIONS:
Overall Officials: Oleg Shapiro, MD, Principal Investigator — State University of New York - Upstate Medical University
Locations (1):
- SUNY Upstate Medical University, Syracuse, New York, United States